CLINICAL TRIAL: NCT05687487
Title: Residual or Recurrent Obstruction After Septal Myectomy in Young Children and Infants With Hypertrophic Cardiomyopathy
Brief Title: Residual or Recurrent Obstruction After Septal Myectomy
Status: Completed | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Jun Yan, Principal Investigator, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2020-I2M-C&T-B-060
Record Dates: First submitted 2023-01-06; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy
Keywords: Septal myectomy; Residual or recurrent obstruction; children and infants; hypertrophic obstructive cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Bites and Stings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to report the outcomes after septal myectomy in young children and infants and identify the mechanisms of residual or recurrent obstruction after surgery. in The main question[s] it aims to answer are:

* What is the early and mid-term results of septal myectomy in young children and infants with severe and extensive obstructive hypertrophic cardiomyopathy (HCM)?
* What are the mechanisms of residual or recurrent obstruction?

Echocardiography and clinical course of children and infants under the age of 14 who underwent septal myectomy for hypertrophic obstructive cardiomyopathy from January 2013 to December 2020 will be followed up.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hypertrophic obstructive cardiomyopathy (HOCM)
* Age young than 14 years
* Patients who have undergone septal myectomy

Exclusion Criteria:

* older than 14 years old;
* secondary left ventricular hypertrophy (LVH) related to subaortic stenosis or aortic stenosis.

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with HOCM who remain severely symptomatic despite medical therapy or have a particularly high resting LVOT gradients (>100mmHg) underwent septal myectomy by the same surgeon Y from January 2013 to December 2020. A total of 56 consecutive children younger than 14 were included. All patients were on Beta blockers therapy and symptomatic.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
death | through study completion, an average of 1 year
  postoperative death during follow-up

SECONDARY OUTCOMES:
recurrent obstruction | through study completion, an average of 1 year
  postoperative recurrent obstruction during follow-up

REFERENCES:
- [Derived] Dong S, Du C, Song J, Dong J, Meng H, Xu H, Sun Y, Zou M, Li S, Yan J. Residual or recurrent obstruction after septal myectomy in young children and infants with hypertrophic cardiomyopathy: cohort study. Int J Surg. 2023 Jun 1;109(6):1699-1707. doi: 10.1097/JS9.0000000000000426. PMID 37165977